CLINICAL TRIAL: NCT05876052
Title: Hypothermic Oxygenated Perfusion To Reduce Tumour Recurrence After Liver Transplantation In Patients With Hepatocarcinoma
Brief Title: HOPE to Reduce Tumour Recurrence After LT In Patients With HCC
Acronym: POTERE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bologna (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); A.O.U. Città della Salute e della Scienza (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Matteo Ravaioli, Professor, Clinical Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POTERE
Record Dates: First submitted 2023-04-21; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Liver Cancer; Tumor Recurrence; Hepatocellular Carcinoma; Liver Transplantation; Ex-vivo Hypothermic Perfusion
MeSH Terms: conditions — Liver Neoplasms; Recurrence; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic oxygenated Perfusion - HOPE (Experimental): Belzer machine perfusion solution at 4°C-10°C in sterile conditions and continuous oxygenation (partial pressure of oxygen=500-600 mmHg) will be used for perfusion, 3000 ml for livers, 1-3 hours.
  Liver perfusion will be performed through the portal vein at a 5 mmHg pressure. Flow, pressure and temperature will be monitored and registered on REDCap software during organ perfusion. Gas analysis of the effluent perfusate (partial pressure O2 and CO2, pH, lactate and glutamate production) will be accomplished every 15 minutes.
  Interventions: Device: Hypothermic oxygenated Perfusion - HOPE
- Static Cold Storage - SCS (No Intervention): Livers undergoing SCS will be stored in sterile organ bags with Belzer or Celsior solution and cooled in ice until transplant.

INTERVENTIONS:
Device: Hypothermic oxygenated Perfusion - HOPE — HOPE will start by flushing the organ at low flow values (30 ml/min) with new oxygenated perfusion fluid during back-table preparation. Organ will be treated with continuous HOPE until transplant. Organ perfusion will be continuously monitored. Minimal perfusion time will be 1 hour for livers.
  Arms: Hypothermic oxygenated Perfusion - HOPE

SUMMARY:
Hypothermic oxygenated ex-situ machine perfusion (HOPE) is a dynamic preservation method that has been developed to reduce the incidence and severity of ischaemia-reperfusion injury and to improve outcomes after liver transplantation. Whit this study Pi and collaborators hypothesize that the application of ex-situ liver perfusion before LT in HCC recipients leads to an optimization of graft function, with a decrease in ischaemia-reperfusion injury and a possible decrease in tumor cell growth. This is multicentre, prospective, two-arm, randomized, controlled, clinical trial, that will will involve patients with HCC candidate to LT. The liver grafts will be randomized in two groups to compare HOPE and static cold storage (SCS) preservation before transplantation. For each group evaluation of clinical outcomes, graft function tests, histologic findings, perfusate, tumor characteristics, and recurrence will be done.

DETAILED DESCRIPTION:
Tumor recurrence after liver transplantation (LT) in patients with hepatocellular carcinoma (HCC) is a major complication leading to decreased long-term survival of patients. However, the mechanisms leading to tumor emergence and growth remain incompletely understood. Several factors, can promote cancer growth or recurrence. Ischemia-reperfusion injury (IRI) has been recognized as an important early driver of microvascular dysfunction resulting in tissue hypoxia and inflammation, which promotes tumor cell growth.

A recent therapeutic strategy used to reduce the incidence and severity of IRI and to improve outcomes after transplantation is ex vivo HOPE. Which allows to redirect anaerobic metabolism to aerobic metabolism under hypothermic conditions, protect grafts from oxidative species-related damage, improve graft function and may potentially reduce cancer recurrence after liver transplantation.

A multicentre, prospective, two-arm, randomized, controlled, clinical trial will be performed; four Italian centres (Bologna, Palermo, Pisa e Torino) will be involved. A total of 192 patients with a history of HCC or active HCC, already present or about to be placed in the liver transplantation waiting list of the four transplantation center will be enroll. The liver grafts will be randomized in two groups to compare HOPE and SCS preservation before transplantation. For each group evaluation of clinical outcomes, graft function tests, histologic findings, perfusate, tumor characteristics, and recurrence will be done during follow up visit; 1-3-6 and 12 months after transplantation.

Livers assigned to HOPE group will be perfused by machine perfusion with cold Belzer solution (4°-10°C) and with continuous oxygenation (partial pressure of oxygen = 500-600 mmHg). Organs will be perfused from the start of the back-table procedure until implantation, without increasing cold ischemia time (CIT).

In the control group livers undergoing SCS will be steeped in cold Celsior or Belzer solutions and stored in ice. Presence of bacterial and/or fungal contamination will be tested by setting up microbiological cultures from the preservation fluid, before and after treatment in both groups.

ELIGIBILITY:
Inclusion Criteria:

* all patients with HCC medical history or active HCC
* Donation after circulatory death (DBD) donor with standard or extended criteria

Exclusion Criteria:

* Living transplantation
* Split Transplantation
* Combined Transplantation
* Donation after cardiac death (DCD)Transplantation
* Re-transplantation
* Patient whose liver graft will undergo ex-vivo machine perfusion for medical decision, regardless the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of liver recurrence | 1 year after LT
  Present/Non present; Diagnosis with abdominal ultrasound and serum tumor markers analysis Date of recurrence and location

SECONDARY OUTCOMES:
Incidence of early allograft disfunction (EAD) | starting 24 hours after LT until 7 days after LT
  Present/Non present;
  Diagnosis with analysis of serum values of :
  Aspartate transaminase (AST), Alanine transaminase (ALT), Bilirubin and International Normalised Ratio (INR)

OTHER OUTCOMES:
Changes in circulating tumor DNA (ctDNA) level | 1 day before LT/ until 12 months after LT
  Blood and tissue samples collection, ctDNA extraction and quantification via Next Generation Sequencing (NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

REFERENCES:
- [Background] Bodzin AS, Lunsford KE, Markovic D, Harlander-Locke MP, Busuttil RW, Agopian VG. Predicting Mortality in Patients Developing Recurrent Hepatocellular Carcinoma After Liver Transplantation: Impact of Treatment Modality and Recurrence Characteristics. Ann Surg. 2017 Jul;266(1):118-125. doi: 10.1097/SLA.0000000000001894. PMID 27433914
- [Background] Boteon YL, Afford SC. Machine perfusion of the liver: Which is the best technique to mitigate ischaemia-reperfusion injury? World J Transplant. 2019 Jan 16;9(1):14-20. doi: 10.5500/wjt.v9.i1.14. PMID 30697517
- [Background] Czigany Z, Schoning W, Ulmer TF, Bednarsch J, Amygdalos I, Cramer T, Rogiers X, Popescu I, Botea F, Fronek J, Kroy D, Koch A, Tacke F, Trautwein C, Tolba RH, Hein M, Koek GH, Dejong CHC, Neumann UP, Lurje G. Hypothermic oxygenated machine perfusion (HOPE) for orthotopic liver transplantation of human liver allografts from extended criteria donors (ECD) in donation after brain death (DBD): a prospective multicentre randomised controlled trial (HOPE ECD-DBD). BMJ Open. 2017 Oct 10;7(10):e017558. doi: 10.1136/bmjopen-2017-017558. PMID 29018070
- [Background] Dutkowski P, Polak WG, Muiesan P, Schlegel A, Verhoeven CJ, Scalera I, DeOliveira ML, Kron P, Clavien PA. First Comparison of Hypothermic Oxygenated PErfusion Versus Static Cold Storage of Human Donation After Cardiac Death Liver Transplants: An International-matched Case Analysis. Ann Surg. 2015 Nov;262(5):764-70; discussion 770-1. doi: 10.1097/SLA.0000000000001473. PMID 26583664
- [Background] Ravaioli M, De Pace V, Angeletti A, Comai G, Vasuri F, Baldassarre M, Maroni L, Odaldi F, Fallani G, Caraceni P, Germinario G, Donadei C, Malvi D, Del Gaudio M, Bertuzzo VR, Siniscalchi A, Ranieri VM, D'Errico A, Pasquinelli G, Morelli MC, Pinna AD, Cescon M, La Manna G. Hypothermic Oxygenated New Machine Perfusion System in Liver and Kidney Transplantation of Extended Criteria Donors:First Italian Clinical Trial. Sci Rep. 2020 Apr 8;10(1):6063. doi: 10.1038/s41598-020-62979-9. PMID 32269237
- [Background] Schlegel A, Muller X, Dutkowski P. Machine perfusion strategies in liver transplantation. Hepatobiliary Surg Nutr. 2019 Oct;8(5):490-501. doi: 10.21037/hbsn.2019.04.04. PMID 31673538
- [Background] Belzer FO, Southard JH. Principles of solid-organ preservation by cold storage. Transplantation. 1988 Apr;45(4):673-6. doi: 10.1097/00007890-198804000-00001. No abstract available. PMID 3282347
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Background] Schlegel A, Muller X, Dutkowski P. Hypothermic Machine Preservation of the Liver: State of the Art. Curr Transplant Rep. 2018;5(1):93-102. doi: 10.1007/s40472-018-0183-z. Epub 2018 Jan 22. PMID 29564206
- [Background] Ravaioli M, Germinario G, Dajti G, Sessa M, Vasuri F, Siniscalchi A, Morelli MC, Serenari M, Del Gaudio M, Zanfi C, Odaldi F, Bertuzzo VR, Maroni L, Laurenzi A, Cescon M. Hypothermic oxygenated perfusion in extended criteria donor liver transplantation-A randomized clinical trial. Am J Transplant. 2022 Oct;22(10):2401-2408. doi: 10.1111/ajt.17115. Epub 2022 Jun 21. PMID 35671067